CLINICAL TRIAL: NCT04045314
Title: Effect of an Emollient Cream Containing 0.5% Cannabidiol and 1% Hemp Oil in the Hydration and Erythema of the Skin
Acronym: Celosia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avicanna Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Av 0001 CeCol
Record Dates: First submitted 2019-07-09; First posted 2019-08-05 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Cosmetics; Eczema
Keywords: CBD; Cosmetics; Dry skin
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Intervention Model Description: This is a prospective, open label, randomized study with passive control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Before-and-after (Experimental): 54 Healthy adults 18 years of age or older at the visit or will receive the first application and will be evaluated according to the objectives defined in the study (short-term data) and to evaluate the long-term effects, two other visits will be made at intervals of 2 weeks to evaluate the impact of topical skin application according to the parameters defined in the study.
  Interventions: Other: Topical moisturizer

INTERVENTIONS:
Other: Topical moisturizer — The investigational product is an intensive emollient cream that is applied topically on the skin and is manufactured by Avicanna Inc. This preparation contains widely used ingredients from mineral and botanical origin aimed at soothing and conditioning the skin as well as improving hydration. The moisturizer also contains 1% hemp oil rich in essential fatty acids and antioxidants as well as 0.5% of CBD with regulatory and conditioning effect on the skin

SUMMARY:
This research seeks to evaluate the short (i.e., after single application) and long-term (i.e., after periodic application) hydrating effect of a topical preparation containing CBD and hemp oil on the skin of the volar forearm as well as the effect on instrumentally measured erythema.

DETAILED DESCRIPTION:
This research seeks to evaluate the short (i.e., after single application) and long-term (i.e., after periodic application) hydrating effect of a topical preparation containing CBD and hemp oil on the skin of the volar forearm as well as the effect on instrumentally measured erythema. Study Design This is a prospective, open label, randomized study with passive control.

Healthy adults will be invited to participate and the general characteristics of the product will be explained, as well as the amount of time that will be required. The individuals that agree to participate will have to read and sign the informed consent, register contact information, and will be scheduled for visit 0 at the research center within 2 to 7 days. During this period, the subject will be told not to use abrasive cleansing products or topical medicines on the volar forearm, not to take more than one shower per day, and not to consume caffeine or alcohol 24 hours before attending the research center.

During the washout period the subject will receive a call to confirm compliance with washout requirements as well as visit 0 schedule. If washout conditions are not met, subject will be reminded to comply and visit will be re-scheduled within 2 to 7 days.

In visit 0 at the research center, contact information, demographic variables and standard anthropometric variables will be recorded. Subsequently, the subject will be given detailed information about the research product and protocol, accompanied by an information leaflet with indications regarding the use of the investigation product as well as recommendations on preferred hygiene regimens.

The subject will be able to review the material in a room under controlled ventilation, temperature, humidity and lighting conditions, where he or she will have to stay for a minimum of 30 minutes. After that, in an adjacent room under the same conditions, the basal characteristics of the skin at the volar forearm and the face will be measured. These are: capacitance, erythema, viscoelasticity and trans-epidermal water-loss (i.e., hour 0) for the volar forearm and erythema for the face. For the face, the bioengineering measurements will be made on at the center of the forehead and for the forearms the anterior surface of the forearms (i.e., volar forearm on both arms) will be used. On the forearms the area to perform measurements will be marked as a 5 by 3 cm rectangle centered at midpoint between the distal wrist crease and the anterior cubital fossa using a skin marker that with removable ink. Additionally, test sites should be uncovered and motionless for at least five minutes before measurement.

Once this process is done, the subject goes back to the waiting room, where a research assistant randomizes the arm using the specially designed field on the platform and explains to the subject how the product must be applied from that moment on (on the face and the forearm). The subject will inspect the product before application and 10 minutes after application will complete a perception survey about the product characteristics and sensation produced on the skin. Afterwards, the subject may leave the room under controlled conditions; however, he or she must return 30 minutes prior to the next measurements.

One hour after the application of the topical product (including 30 minutes of acclimatization in the room under controlled conditions), a new measurement of the capacitance, erythema, viscoelasticity and trans-epidermal water-loss is made. This procedure is repeated after 3 hours (including 30 minutes of acclimatization in the room under controlled conditions). Once the last measurement is made the subject completes the last part of the survey and is given a vessel containing the investigational product and instructions regarding its usage will be reinforced. Additionally, schedule for next visit will be determined at this time.

The subject must apply the product according to the indications and keep a journal of the applications. Additionally, the subject must refrain from using other topical products on the volar forearm or systemic products that may alter the skin conditions. Furthermore, there will be a follow-up call to remind the participant to comply with the requirements and confirm schedule next visit.

Two weeks after visit 0, the subject will return to the research center, where a new measurement of the capacitance, erythema, viscoelasticity and trans-epidermal water-loss is made. This procedure is repeated by the 4th week, additionally, the subject will answer the last part of the perception survey in this visit. Once this is completed the product application phase will be terminated and the amount of remaining product as well as any significant journal entries will be registered at this point.

Throughout the study there will be tolerance and safety monitoring in every visit and follow-up call, as follows: Upon first application of the investigational product there will be an observation of the subject during a 15-minute period done by the research staff, a physician will be available to assess any possible allergic reaction or significant irritation.

The research staff will examine the application site of the research product to find potential local reactions and will ask about any systemic symptom. If no adverse reactions occur, the information will be recorded. Similarly, if any adverse reaction, systemic reaction or adverse event occurs it will be recorded and the physician will take the necessary measures to ensure subject safety according to his expert judgement and initiate event reporting according to applicable regulation. Finally, in every phone call made by the call center, adherence and tolerance questions will be made and recorded.

At the 5th week, the subject will receive a final follow-up call to record any events that might have appeared after removing the product, thus ending follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

* Adult (i.e., over 18 years old) men or women.
* Dry skin (i.e., Modified Kligman test >0)
* Accepts and signs the informed consent.

Exclusion Criteria

* Pregnant or breast-feeding women
* Subjects with a chronic disease that requires medication
* Subjects with known diagnosis of cancer
* Smoking habit or alcohol consumption habit (i.e., once a day or more)
* Recreational o medicinal cannabinoid use
* Skin diseases (i.e., diseases that require care of a dermatologist)
* Current medication uses such as: Immunomodulators, antibiotics, corticoids or retinoids
* Hypersensitivity to any component of the research product
* Involvement in other clinical or cosmetic studies in the last 6 months
* Recent exposure to sun causing sun tanning (i.e., as reported by the subject causing discomfort or change in the usual appearance of the skin)
* Permanent decoration of the skin in the test area

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect on hydration of a single application of the topical preparation on facial skin | 1 and 3 hours
  1. Evaluate the effect on hydration of a single application of the topical preparation on the skin of the volar forearm, through the direct measurement of its electrical properties as an indicator of water content at 1 and 3 hours
Evaluate the effect on Hydration of periodic application of the topical preparation on facial skin | 2 and 4 weeks
  2. Evaluate the effect on hydration of periodic application of the topical preparation on facial skin, through the direct measurement of its electrical properties as an indicator of water content at 2 and 4 weeks.

SECONDARY OUTCOMES:
Evaluate the short-term change in instrumentally assessed erythema | Up to 3 hours
  Evaluate the short-term change in instrumentally assessed erythema (i.e., 1 and 3 hours), through the direct measurement of skin biochromophores at the face and the volar forearm.
Evaluate the long-term change in instrumentally assessed erythema | 4 weeks
  Evaluate the long-term change in instrumentally assessed erythema (i.e., 2 and 4 weeks), through the direct measurement of skin biochromophores at the face and the volar forearm.
Evaluate the short-term effect of this topical preparation on the viscoelastic properties of the skin | 3 hours
  Evaluate the short-term effect (i.e., 1 and 3 hours) of this topical preparation on the viscoelastic properties of the skin, through the direct measurement of its response to physical deformation by suction.
Evaluate the long-term effect of this topical preparation on the viscoelastic properties of the skin | 4 weeks
  Evaluate the long-term effect (i.e., 2 and 4 weeks) of this topical preparation on the viscoelastic properties of the skin, through the direct measurement of its response to physical deformation by suction.
Evaluate the short-term effect of this topical preparation on the skin functional properties | 3 hours
  Evaluate the short-term effect (i.e., 1 and 3 hours) of this topical preparation on the skin functional properties, through the measurement of trans-epidermal water loss.
Evaluate the long-term effect of this topical preparation on the skin functional properties | 4 weeks
  Evaluate the long-term effect (i.e., 2 and 4 weeks) of this topical preparation on the skin functional properties, through the measurement of trans-epidermal water loss.
Evaluate the short and long-term appearance of evaluator assessed irritation | 4 weeks
  Evaluate the short and long-term appearance of evaluator assessed irritation by visual scoring (i.e., 0 hours, 1 hours and 4 weeks).
  Perceived skinfeel attributes of creams and lotions (appearance, rub-in, absorption, appearance of skin, immediate and delayed after-feel) have been evaluated using a trained descriptive panel. In previously published studies researchers used the skinfeel spectrum descriptive analysis method to characterize skin care products. They used strict protocols for manipulation and precisely defined terms to describe the qualitative properties and their relative intensities in each product. The evaluation process was divided into four categories: pick-up (i.e., firmness, stickiness, cohesiveness, peaking); rub-out (i.e., wetness, spreadability, thickness, absorbency); residual feel; and appearance, immediate and after 20 minutes (i.e., glossy, sticky, slippery, oily, waxy, greasy)
Evaluate the short and long-term emollient effect and acceptance | 4 weeks
  Evaluate the short and long-term emollient effect and acceptance of this topical preparation, through the application of a perception survey (i.e., 0 hours, 1 hours and 4 weeks).
  Perceived skinfeel attributes of creams and lotions (appearance, rub-in, absorption, appearance of skin, immediate and delayed after-feel) have been evaluated using a trained descriptive panel. In previously published studies researchers used the skinfeel spectrum descriptive analysis method to characterize skin care products. They used strict protocols for manipulation and precisely defined terms to describe the qualitative properties and their relative intensities in each product. The evaluation process was divided into four categories: pick-up (i.e., firmness, stickiness, cohesiveness, peaking); rub-out (i.e., wetness, spreadability, thickness, absorbency); residual feel; and appearance, immediate and after 20 minutes (i.e., glossy, sticky, slippery, oily, waxy, greasy)

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Granados, MD., MSc., Principal Investigator — Centro de Atencion e Investigacion Medica
Locations (1):
- VITA, Chía, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapoor S, Saraf S. Assessment of viscoelasticity and hydration effect of herbal moisturizers using bioengineering techniques. Pharmacogn Mag. 2010 Oct;6(24):298-304. doi: 10.4103/0973-1296.71797. PMID 21120032
- [Background] Fleck O, Vejrup-Hansen R, Watson A, Carr AM, Nielsen O, Holmberg C. Spd1 accumulation causes genome instability independently of ribonucleotide reductase activity but functions to protect the genome when deoxynucleotide pools are elevated. J Cell Sci. 2013 Nov 1;126(Pt 21):4985-94. doi: 10.1242/jcs.132837. Epub 2013 Aug 28. PMID 23986475
- [Background] Wickett RR, Damjanovic B. Quantitation of 24-Hour Moisturization by Electrical Measurements of Skin Hydration. J Wound Ostomy Continence Nurs. 2017 Sep/Oct;44(5):487-491. doi: 10.1097/WON.0000000000000363. PMID 28877115
- [Background] Biro T, Toth BI, Hasko G, Paus R, Pacher P. The endocannabinoid system of the skin in health and disease: novel perspectives and therapeutic opportunities. Trends Pharmacol Sci. 2009 Aug;30(8):411-20. doi: 10.1016/j.tips.2009.05.004. Epub 2009 Jul 14. PMID 19608284
- [Background] Kupczyk P, Reich A, Szepietowski JC. Cannabinoid system in the skin - a possible target for future therapies in dermatology. Exp Dermatol. 2009 Aug;18(8):669-79. doi: 10.1111/j.1600-0625.2009.00923.x. PMID 19664006
- [Background] Citti C, Pacchetti B, Vandelli MA, Forni F, Cannazza G. Analysis of cannabinoids in commercial hemp seed oil and decarboxylation kinetics studies of cannabidiolic acid (CBDA). J Pharm Biomed Anal. 2018 Feb 5;149:532-540. doi: 10.1016/j.jpba.2017.11.044. Epub 2017 Nov 20. PMID 29182999
- [Background] Mikulcova V, Kasparkova V, Humpolicek P, Bunkova L. Formulation, Characterization and Properties of Hemp Seed Oil and Its Emulsions. Molecules. 2017 Apr 27;22(5):700. doi: 10.3390/molecules22050700. PMID 28448475
- [Background] Eccles M, Grimshaw J, Campbell M, Ramsay C. Research designs for studies evaluating the effectiveness of change and improvement strategies. Qual Saf Health Care. 2003 Feb;12(1):47-52. doi: 10.1136/qhc.12.1.47. PMID 12571345
- [Background] Rawlings AV, Canestrari DA, Dobkowski B. Moisturizer technology versus clinical performance. Dermatol Ther. 2004;17 Suppl 1:49-56. doi: 10.1111/j.1396-0296.2004.04s1006.x. PMID 14728699
- [Background] Petry T, Bury D, Fautz R, Hauser M, Huber B, Markowetz A, Mishra S, Rettinger K, Schuh W, Teichert T. Review of data on the dermal penetration of mineral oils and waxes used in cosmetic applications. Toxicol Lett. 2017 Oct 5;280:70-78. doi: 10.1016/j.toxlet.2017.07.899. Epub 2017 Aug 5. PMID 28789996
- [Background] Reuter J, Merfort I, Schempp CM. Botanicals in dermatology: an evidence-based review. Am J Clin Dermatol. 2010;11(4):247-67. doi: 10.2165/11533220-000000000-00000. PMID 20509719
- [Background] Iffland K, Grotenhermen F. An Update on Safety and Side Effects of Cannabidiol: A Review of Clinical Data and Relevant Animal Studies. Cannabis Cannabinoid Res. 2017 Jun 1;2(1):139-154. doi: 10.1089/can.2016.0034. eCollection 2017. PMID 28861514
- [Background] Graham JE, Karmarkar AM, Ottenbacher KJ. Small sample research designs for evidence-based rehabilitation: issues and methods. Arch Phys Med Rehabil. 2012 Aug;93(8 Suppl):S111-6. doi: 10.1016/j.apmr.2011.12.017. Epub 2012 May 8. PMID 22580169
- [Background] Darlenski R, Sassning S, Tsankov N, Fluhr JW. Non-invasive in vivo methods for investigation of the skin barrier physical properties. Eur J Pharm Biopharm. 2009 Jun;72(2):295-303. doi: 10.1016/j.ejpb.2008.11.013. Epub 2008 Dec 11. PMID 19118626
- [Background] Fluhr JW, Darlenski R, Angelova-Fischer I, Tsankov N, Basketter D. Skin irritation and sensitization: mechanisms and new approaches for risk assessment. 1. Skin irritation. Skin Pharmacol Physiol. 2008;21(3):124-35. doi: 10.1159/000131077. Epub 2008 Jun 3. PMID 18523410
- [Background] Fluhr JW, Kuss O, Diepgen T, Lazzerini S, Pelosi A, Gloor M, Berardesca E. Testing for irritation with a multifactorial approach: comparison of eight non-invasive measuring techniques on five different irritation types. Br J Dermatol. 2001 Nov;145(5):696-703. doi: 10.1046/j.1365-2133.2001.04431.x. PMID 11736891
- [Background] Nedelec B, Forget NJ, Hurtubise T, Cimino S, de Muszka F, Legault A, Liu WL, de Oliveira A, Calva V, Correa JA. Skin characteristics: normative data for elasticity, erythema, melanin, and thickness at 16 different anatomical locations. Skin Res Technol. 2016 Aug;22(3):263-75. doi: 10.1111/srt.12256. Epub 2015 Sep 1. PMID 26333046
- [Background] Edwards C, Marks R. Evaluation of biomechanical properties of human skin. Clin Dermatol. 1995 Jul-Aug;13(4):375-80. doi: 10.1016/0738-081x(95)00078-t. PMID 8665446
- [Background] Jemec GB, Wulf HC. The plastic sing effect of moisturizers on human skin in vivo: a measure of moisturizing potency? Skin Res Technol. 1998 May;4(2):88-93. doi: 10.1111/j.1600-0846.1998.tb00092.x. PMID 27332105
- [Background] Dobrev H. Use of Cutometer to assess epidermal hydration. Skin Res Technol. 2000 Nov;6(4):239-244. doi: 10.1034/j.1600-0846.2000.006004239.x. PMID 11428963
- [Background] Loden M. The clinical benefit of moisturizers. J Eur Acad Dermatol Venereol. 2005 Nov;19(6):672-88; quiz 686-7. doi: 10.1111/j.1468-3083.2005.01326.x. PMID 16268870
- [Background] Lukic M, Jaksic I, Krstonosic V, Cekic N, Savic S. A combined approach in characterization of an effective w/o hand cream: the influence of emollient on textural, sensorial and in vivo skin performance. Int J Cosmet Sci. 2012 Apr;34(2):140-9. doi: 10.1111/j.1468-2494.2011.00693.x. Epub 2011 Dec 6. PMID 22085371